CLINICAL TRIAL: NCT05249959
Title: Consolidation With ADCT-402 (Loncastuximab Tesirine) After a Short Course of Immunochemotherapy: a Phase II Study in BTKi-treated (or BTKi Intolerant) Relapsed/Refractory (R/R) Mantle Cell Lymphoma (MCL) Patients
Brief Title: Consolidation With Loncastuximab Tesirine After a Short Course of Immunochemotherapy in BTKi-treated (or Intolerant) Relapsed/Refractory Mantle Cell Lymphoma Patients.
Acronym: FIL_COLUMN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_COLUMN
Record Dates: First submitted 2022-02-03; First posted 2022-02-22 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Relapsed Mantle Cell Lymphoma; Refractory Mantle Cell Lymphoma
Keywords: Relapsed/Refractory Mantle Cell Lymphoma (MCL); ADCT-402 (loncastuximab tesirine); BTKi (Bruton Tyrosine Kinase inhibitors) - treated; BTKi (Bruton Tyrosine Kinase inhibitors) intolerant
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — loncastuximab tesirine; Cytarabine

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, phase II single arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Consolidation with ADCT-402 (loncastuximab tesirine) after a short course of immunochemotherapy (Experimental): R/R MCL after one, two, three or four lines of treatment including BTKi treatment (or BTKi intolerant), with complete response (CR) or partial response (PR) or with stable disease (SD) after salvage immunochemotherapy (R-BAC, Rituximab - Bendamustine, Ara-C x 2 cycles) will undergo consolidation with loncastuximab tesirine. A patient with CR, PR or SD after one R-BAC course, which is unable to undergo a second course due to toxicity to chemotherapy, can be considered to proceed for consolidation.
  Interventions: Drug: Consolidation with ADCT-402 (loncastuximab tesirine) after salvage immunochemotherapy at standard dose (R-BAC, Rituximab - Bendamustine, Ara-C)); Drug: Consolidation with ADCT-402 (loncastuximab tesirine) after salvage immunochemotherapy at reduced dose (R-BAC, Rituximab - Bendamustine, Ara-C)

INTERVENTIONS:
Drug: Consolidation with ADCT-402 (loncastuximab tesirine) after salvage immunochemotherapy at standard dose (R-BAC, Rituximab - Bendamustine, Ara-C)) — Standard Induction phase (cycle 1-2 of R-BAC every 28 days according to the following schedule):
  * Rituximab 375 mg/m2 i.v. Day 1
  * Bendamustine 70 mg/m2, Days 2 and 3
  * Cytarabine 500 mg/m2, Day 2-4
  After restaging at the End of Induction (EOI) patients with CR (complete response), PR (partial response) or SD (stable disease) will receive:
  CONSOLIDATION PHASE:
  * 2 infusions of loncastuximab tesirine at a dose of 150 microgram/kg every three weeks followed by
  * 2 infusions of loncastuximab tesirine at a dose of 75 microgram/kg every three weeks
Drug: Consolidation with ADCT-402 (loncastuximab tesirine) after salvage immunochemotherapy at reduced dose (R-BAC, Rituximab - Bendamustine, Ara-C) — Reduced Induction phase (cycle 1-2 with two different schedules for patients deemed FRAIL or UNFIT for standard induction therapy,based on protocol dose and as per medical judgment are allowed).
  * Rituximab 375 mg/m2 i.v. Day 1
  * Bendamustine 70 mg/m2, Days 2 and 3
  * Cytarabine 500 mg/m2, Day 2 and 3
  or
  * Rituximab 375 mg/m2 i.v. Day 1
  * Bendamustine 100 mg, Days 2 and 3
  * Cytarabine 500 mg, Day 2 and 3
  After restaging at the End of Induction (EOI) patients with CR (complete response), PR (partial response) or SD (stable disease) will receive:
  CONSOLIDATION PHASE:
  * 2 infusions of loncastuximab tesirine at a dose of 150 microgram/kg every three weeks followed by
  * 2 infusions of loncastuximab tesirine at a dose of 75 microgram/kg every three weeks

SUMMARY:
This is a prospective, phase 2, multicenter, open-label, single-arm study. Primary objective is to assess the efficacy of loncastuximab tesirine given as consolidation therapy after salvage immunochemotherapy in BTKi (Bruton Tyrosine Kinase inhibitors) -treated (or BTKi intolerant) R/R (Relapse or Refractory) MCL (Mantle Cell Lymphoma) patients. The sponsor of this clinical trial is Fondazione Italiana Linfomi - ETS (FIL ETS).

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, open-label, single-arm study of the efficacy and safety of loncastuximab tesirine given as consolidation therapy after salvage immunochemotherapy in BTKi-treated (or BTKi intolerant) R/R MCL patients.

Primary Objective:

- To assess the efficacy of a consolidation with loncastuximab tesirine following salvage immunochemotherapy (2 courses of Rituximab-Bendamustine-Cytarabine, R-BAC) in Bruton Tyrosine Kinase inhibitors (BTKi) treated (or BTKi intolerant) relapsed/refractory (R/R) Mantle Cell Lymphomas (MCL).

Secondary Objectives:

* To evaluate the safety profile of loncastuximab tesirine consolidation.
* To assess the rate of Minimal Residual Disease (MRD) negativity after loncastuximab tesirine consolidation.

R/R MCL patients after one, two, three or four lines of treatment including BTKi treatment (or BTKi intolerant), with complete response (CR) or partial response (PR) or with stable disease (SD) after salvage immunochemotherapy (R-BAC x 2, Rituximab - Bendamustine, Cytarabine) will undergo consolidation with loncastuximab tesirine. A patient with CR, PR or SD after one R-BAC course, which is unable to undergo a second course due to toxicity to chemotherapy, can be considered to proceed for consolidation.

After checking inclusion and exclusion criteria and signing written informed consent, patients will be enrolled in the study, and the system will assign them an alphanumeric code that will identify the patient in every study procedure.

Efficacy parameters will be evaluated according to the Lugano 2014 Classification.

Toxicity parameters will be evaluated according to the definitions of the current version of the NCI (National Cancer Institute) CTCAE (Common Terminology Criteria for Adverse Events) criteria.

After treatment discontinuation, both in the case the protocol treatment was fully administered and in the case of an early discontinuation, patients will be followed-up according to clinical practice timeline and procedures, and information on patient status (progression/relapse, alive/dead, lost to follow-up) will be collected till the end of the study (LPLV), planned 36 months after the start of treatment of the last patient enrolled in the study. In case of progression/relapse during follow-up, the patients will be then followed-up for survival till the study end.

49 patients will be enrolled in the study.

The anticipated study dates are:

* Total accrual period: 48 months
* Last patient last visit (LPLV): 36 months after the start of treatment of the last patient enrolled.

The study will include a period of screening up to 21 days, a period of treatment of up to 22 weeks and a follow-up period with visits every 4-8 weeks for the first year after study entry and then every 8-12 weeks for at least 2 years.

Treatment includes a period of induction with 2 cycles of 28 days with R-BAC (=8 weeks) + two/four weeks for restaging + 4 doses of loncastuximab tesirine every 21 days (=12 weeks), i.e., a total period of 22 weeks, for patients who achieved CR, PR or SD after salvage immunochemotherapy. A follow-up period with visits every 4-8 weeks for the first year after study entry and then every 8-12 weeks for at least to 2 years.

For the study is also planned an extended follow-up after the end of the study requiring participating sites to provide only information on patient status (alive, dead, lost to follow-up) and to record possible events occurred after the end of the study, including diagnosis of second neoplasia and long-term toxicity for additional 2 years after the end of the study.

Disease evaluation will be performed initially (Baseline Assessment), after the beginning of treatment with R-BAC (End of Induction), at the end of loncastuximab tesirine consolidation phase (End of Treatment) and then every 6 months during the follow-up period.

Non-responder, relapsing or progressive patients will be treated according to best clinical practice.

Treatment schedule:

Standard Induction phase:

2 courses of R-BAC every 28 days according to the following schedule

* Rituximab 375 mg/m2 i.v. Day 1
* Bendamustine 70 mg/m2, Days 2 and 3
* Cytarabine 500 mg/m2, Day 2-4

Reduced Induction phase:

For patients deemed FRAIL or UNFIT for standard induction therapy (based on protocol dose and as per medical judgment), reduced R-BAC options may be considered. For patients > 80 years old the reduced induction schedule is recommended.

Two different schedules will be allowed

Cycle 1-2

* Rituximab 375 mg/m2 i.v. Day 1
* Bendamustine 70 mg/m2, Days 2 and 3
* Cytarabine 500 mg/m2, Day 2 and 3

or

Cycle 1-2

* Rituximab 375 mg/m2 i.v. Day 1
* Bendamustine 100 mg, Days 2 and 3
* Cytarabine 500 mg, Day 2 and 3

An optional pre-phase with steroid (prednisone 1 mg/kg/day, maximum of 7 days before starting induction phase) and/or single dose of Vincristine (up to 2 mg total) was allowed.

After restaging at the End of Induction (EOI) patients with CR, PR or SD will receive:

CONSOLIDATION PHASE:

* 2 infusions of loncastuximab tesirine at a dose of 150 microgram/kg* every three weeks followed by
* 2 infusions of loncastuximab tesirine at a dose of 75 microgram/kg* every three weeks

  * (For patients with BMI> 35 dose will be calculated based on adjusted weight). Patients will undergo initial staging with CT (Computed Tomography) scan, PET (18F-FDG Positron Emission Tomography)/PET-CT scan and bone marrow (BM) biopsy. Patients will be fully restaged after induction (EOI), after loncastuximab tesirine consolidation (EOT) and then every six months only with CT-scan.

Tumour re-biopsy will be performed only if clinically indicated. Bone Marrow (BM) and Peripheral Blood (PB) samples for MRD evaluation purposes will be taken at the same time points when CT-scan is done (to be performed centrally at certified Euro-MRD academic laboratories, according to Euro-MRD guidelines).

Response to treatment will be evaluated according to the Lugano 2014 criteria. Based on published results we considered the expected 12-month PFS with available treatments to be <20%; we hypothesized that, in this setting of patients, a consolidation with loncastuximab tesirine (ADCT-402) may increase the expected 12-month PFS to ≥40% According to one arm non-parametric survival provided by SWOG (Southwest Oncology Group-NCI), with an alpha error (one sided) equal to 0.05, a beta error equal to 0.10, 2-years of accrual and a minimum of 3 year of follow-up, the required sample size consist of 49 patients who start treatment after screening phase. The lower limit of the 90% confidence interval (according to 1-sided alpha error of 0.05) of the 12-month PFS must be higher than the null hypothesis of 0.20 to conclude that the new treatment is promising for a subsequent phase III study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented diagnosis of MCL as defined in the 2017 edition of the World Health Organization (WHO) classification
* Age ≥ 18 and < 85 years
* Relapsed/Refractory disease after one, two, three or four lines of treatment
* Bendamustine-naive or relapsed after at least one year after the last cycle of a bendamustine-containing regimen
* Previous treatment with BTKi (Bruton Tyrosine Kinase inhibitors) monotherapy or BTKi containing regimens with R/R disease; and/or patients who discontinued BTKi monotherapy or BTKi containing regimens for adverse events and have active disease necessitating treatment.
* Previous treatment with any anti-CD19 agents is allowed (included CAR-T treatment) If previous anti-CD19 treatment has occurred, tissue CD19 expression must be assessed by histology or flow cytometry
* Venetoclax treated patients are allowed.
* Stem cell transplant eligible patients are allowed.
* Measurable nodal or extranodal disease ≥ 1.5 cm in longest diameter, and measurable in 2 perpendicular dimensions. Note: Patients with bone marrow involvement only are eligible. In case of bone marrow infiltration only, bone marrow aspiration and biopsy are mandatory for all staging evaluations
* ECOG (Eastern Cooperative Oncology Group)/WHO (World Health Organization) performance status ≤ 2 (unless MCL-related)
* The following laboratory values at screening (unless due to bone marrow involvement by lymphoma):

  * Absolute Neutrophil count (ANC) > 1.0×109/L
  * Platelet count ≥ 75.000/mm3
  * Creatinine clearance ≥ 40 mL/min (Cockcroft-Gault formula)
  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 x ULN (upper limit of normal)
  * Bilirubin ≤ 1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non- hepatic origin)
* Subject understands and voluntarily signs an informed consent form approved by an Independent Ethics Committee (IEC), prior to the initiation of any screening or study-specific procedures.
* Subject must be able to adhere to the study visit schedule and other protocol requirements.
* Life expectancy ≥ 3 months.
* Women of childbearing potential (WOCBP) and men must agree to use effective contraception if sexually active.This applies for the time period between signing of the informed consent form and at least 10 months after last loncastuximab tesirine (ADCT-402) dose. Men with female partners who are of childbearing potential must agree to use effective contraception if sexually active. This applies for the time period between signing of the informed consent form and at least 7 months after last loncastuximab tesirine (ADCT-402) dose.

Exclusion Criteria:

* Subjects who have received a bendamustine containing regimen and relapsed less than one year after the end of treatment.
* Known history of hypersensitivity to human antibodies.
* Allogenic stem cell transplant within 6 months prior to start of first study drug.
* Allogenic stem cell transplant with active / uncontrolled graft-versus-host disease.
* Previous treatment with CD19 targeting agents.
* More than four lines of previous treatment (autologous stem cell transplant performed as part of consolidation to a previous line of therapy should not be considered as a line of therapy).
* Active second malignancy in the last three years other than non-melanoma skin cancers, non-metastatic prostate cancer, in situ cervical cancer, ductal or lobular carcinoma in situ of the breast, or any other tumor that the Sponsor and Coordinating Investigator agree and document should not be considered preclusive to participate in the study.
* Major surgery or any anticancer therapy including chemotherapy, immunotherapy, radiotherapy, investigational therapy, including targeted small molecule agents within 14 days prior to start of study drug (R-BAC). A shorter interval in special settings must be approved by the Sponsor and/or Investigator.
* Cardiovascular disease (NYHA, New York Heart Association, class ≥2).
* Significant history of neurologic, psychiatric, endocrinological, metabolic, immunologic, or hepatic disease that would preclude participation in the study or compromise ability to give informed consent.
* Evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

  * Uncontrolled and/or active systemic infection (viral including COVID 19, bacterial or fungal);
  * Chronic or acute hepatitis B (HBV) or hepatitis C (HCV) requiring treatment. Note:

subjects with serologic evidence of prior vaccination to HBV (i.e., HBsAg negative, HBsAb positive and HBcAb negative) or positive HBcAb from previous infection or intravenous immunoglobulins (IVIG) may participate; inactive carriers (HBsAg positive with undetectable HBV DNA) are eligible. Patients with presence of HCV antibody are eligible only if PCR results (polimerase chain reaction) negative for HCV RNA.

* HIV seropositivity.
* Lymphoma with active CNS (central nervous system) involvement at the time of screening, including leptomeningeal disease.
* Congenital long QT syndrome or a corrected QTcF interval of >480 msec at screening (unless secondary to pacemaker or bundle branch block).
* Any other significant medical illness, abnormality, or condition that would, in the Investigator's judgment, make the patient inappropriate for study participation or put the patient at risk.
* If female, the patient is pregnant or breast-feeding.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2026-03-21 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | The primary endpoint will be assessed from the beginning of the study up to 36 months.
  The length of time during and after the treatment that patients live with the disease, but it does not get worse. Progression-Free Survival (PFS) will be defined from the date of enrollment and the first documentation of recurrence, progression or death from any cause. Responding patients and patients who are lost to follow up will be censored at their last assessment date. PFS will be assessed on an ITT (Intention to Treat) basis.

SECONDARY OUTCOMES:
Overall Survival (OS) | The endpoint will be assessed from the beginning of the study up to 36 months
  The percentage of patients alive. The endpoint is defined as the time between the start of treatment until death from any cause; patients who are lost at follow up will be censored at their last assessment date. Analysis will be performed on an ITT (Intention to Treat) basis.
Overall Response Rate (ORR) | The endpoint will be assessed from the beginning of the study therapy up to 6 months
  Overall response rate (ORR) is defined as the proportion of patients who have a complete response (CR), or partial response (PR) or stable disease (SD) to therapy.
  Overall Response Rate (ORR) will be defined according to the Lugano 2014 criteria. The best overall response will be defined as the best response between the date of beginning of therapy and the last restaging. Patients without response assessment (due to whatever reason) will be considered as non-responders.
Duration of Response (DOR) | The endpoint will be assessed from the beginning of the study therapy up to 36 months
  The length of time that the disease continues to respond to treatment without growing or spreading.
  It is also defined as the time from the first documentation of tumor response (CR/PR) to disease progression or death according to Lugano 2014 Criteria. Analysis will be performed on an ITT (Intention to Treat) basis.
Event-Free Survival (EFS) | The endpoint will be assessed from the beginning of the study therapy up to 36 months
  The measure of time after treatment that patients have not have cancer come back or get worse.
  It is also defined as the time from start of treatment to disease progression, death, or discontinuation of treatment for any reason (e.g. toxicity, patient preference), or initiation of a new treatment without documented progression. Analysis will be performed on an ITT (Intention to Treat) basis.
MRD (Minimal Residual Disease) negativity rate | The endpoint will be assessed from the beginning of the study therapy up to 18 months
  The percentage of patients with negative Minimal Residual Disease (MRD) after induction treatment, at the end of consolidation with loncastuximab tesirine and after 6 and 12 months after the end of consolidation.
Rate of Adverse Events | The endpoint will be assessed from the beginning of the study therapy up to 36 months
  Percentage of toxicities. Any grade III or higher toxicities will be recorded and classified according to the definitions of the current version of the NCI Common Terminology Criteria for Adverse Events (CTCAE).
Rate of conversion from partial response (PR) to complete response (CR) | The endpoint will be assessed from the beginning of the study therapy up to 6 months
  Percentage of patients that turn from a partial respons to a complete response. This endpoint will be assessed by comparing responses prior to and after loncastuximab tesirine
Rate of conversion from stable disease (SD) to complete response (CR) and partial response (PR) | The endpoint will be assessed from the beginning of the study therapy up to 6 months
  Percentage of patients that turn from a stable disease to a complete response and partial response .This endpoint will be assessed by comparing responses prior to and after loncastuximab tesirine

CONTACTS AND LOCATIONS:
Overall Officials: Marco Ladetto, Principal Investigator — S.C. Ematologia - A.S.O. "SS Antonio e Biagio e Cesare Arrigo" di Alessandria
Locations (21):
- Italy (21):
  - ASST Spedali Civili di Brescia, Brescia, Italy
  - S.C. Ematologia - A.S.O. "SS Antonio e Biagio e Cesare Arrigo", Alessandria
  - S.C. di Ematologia - A.O. S. Croce e Carle, Cuneo
  - Unità funzionale di Ematologia - Azienda Ospedaliera Universitaria Careggi, Florence
  - Ematologia - Ospedale Policlinico San Martino S.S.R.L. - IRCCS per l'Oncologia, Genova
  - Ematologia - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Milan
  - S.C. Ematologia - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - UOC Ematologia Oncologica - Istituto Nazionale Tumori - IRCCS Fondazione G. Pascale, Napoli
  - SCDU Ematologia - AOU Maggiore della Carità di Novara, Novara
  - Divisione di Ematologia - A.O. Ospedali Riuniti Villa Sofia-Cervello, Palermo
  - Divisione di Ematologia - IRCCS Policlinico S. Matteo di Pavia, Pavia
  - Ematologia - Ospedale delle Croci, Ravenna
  - Ematologia - Azienda Unitа Sanitaria Locale-IRCCS - Arcispedale Santa Maria Nuova, Reggio Emilia
  - U.O. di Ematologia - Ospedale degli Infermi di Rimini, Rimini
  - Dipartimento di Medicina Traslazionale e di Precisione - Policlinico Umberto I - Università "La Sapienza" Istituto Ematologia, Roma
  - U.O. Ematologia - Istituto Clinico Humanitas, Rozzano
  - S.C. Ematologia Universitaria - A.O.U. Città della Salute e della Scienza di Torino, Torino
  - S.C di Ematologia - Ospedale Ca Foncello, Treviso
  - U.O.C Ematologia e Trapianto - A.O. C. Panico, Tricase
  - SC Ematologia - Azienda Sanitaria Universitaria Giuliano Isontina (ASUGI), Trieste
  - U.O. Ematologia - AOU Integrata di Verona, Verona